CLINICAL TRIAL: NCT03717753
Title: The Association Between a Comprehensive Multimodal Pathway And Pain 0-48 Hours After Arthroscopic Rotator Cuff Repair: A Before-and After Study
Brief Title: Rotator Cuff Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0814
Record Dates: First submitted 2018-09-12; First posted 2018-10-24 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before Group (No Intervention): We plan to have 70 patients studied prior to initiation of a pathway.
- After Group (Experimental): We plan to have 70 patients studied after initiation of a pathway.
  Interventions: Other: Pathway

INTERVENTIONS:
Other: Pathway — The study team emphasizes that all components of the pathway are considered standard of care at this institution. The objective of this study is to ensure that the study patients assigned to the pathway will receive these standard of care components. Both groups will receive identical postoperative follow-up.
  Arms: After Group

SUMMARY:
Rotator cuff surgery is mostly performed on an outpatient basis, and many patients still experience moderate to severe pain after surgery, despite the use of regional anesthesia and opioids. The specific aim is to determine whether a comprehensive pathway that includes a well-defined regional technique and multimodal analgesia will reduce the worst pain with movement 0-48 hours after block placement compared to the current standard practice. This is a 'before and after' study. We plan to have 70 patients studied prior to initiation of a pathway, and 70 patients studied after initiation of a pathway. Both groups will receive identical postoperative follow-up.

DETAILED DESCRIPTION:
Previous study in shoulder arthroplasty patients demonstrated low pain scores and minimal intravenous opioid use when utilizing a clinical pathway that included peripheral nerve block and preemptive non-opioid analgesia (Goon et al. 2014). These surgeries were done as inpatient and patients had availability of intravenous opioids. Assessment of the current approach to managing rotator cuff repairs demonstrated an average worst pain score after surgery of 7.0, SD 2.1 (Kahn) which is often categorized as "severe" pain. Given that most rotator cuff repairs are done as outpatients, it is important to develop a clinical pathway that mitigates the worst pain experienced after surgery. With outpatient surgery, there are obvious limitations regarding availability of rescue pain medications. Therefore, the pathway needs to emphasize patient education and strategies to reduce the pain as peripheral nerve block subsides. Given these issues, we believe there is an advantage to prolonging the analgesia from the nerve block (Rosenfeld et al. 2016, Yadeau et al. 2016, Kahn) and educating patients regarding the importance of preemptive analgesia and when to take opioid medications. This study will evaluate whether the clinical pathway might mitigate the worst pain after surgery that occurs with the current standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory rotator cuff patients with participating surgeons.

Includes the following concomitant procedures:

* Arthroscopic SLAP (Superior Labrum Anterior and Posterior) repair
* Arthroscopic Stabilization
* Arthroscopic AC (Acromioclavicular) resection
* Arthroscopic SAD (Sub-Acromial Decompression)
* Arthroscopic or mini open biceps tenodesis
* Age 18-80

Exclusion Criteria:

* chronic pain history (defined as use of opioids > 3 months or current gabapentinoids for pain)
* open surgery (but sub pectoralis mini open biceps tenodesis is not excluded)
* revision surgery
* kidney disease (GFR < 60 ml/min/1.73 m2 for 3 months or more)
* liver disease (transaminitis, cirrhosis, hepatitis, hypoalbuminemia, coagulopathy)
* planned avoidance of regional anesthesia
* any contraindication to or patient refusal of any component in the pathway
* Non-English speakers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques YaDeau, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital of Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] YaDeau JT, Soffin EM, Tseng A, Zhong H, Dines DM, Dines JS, Gordon MA, Lee BH, Kumar K, Kahn RL, Kirksey MA, Schweitzer AA, Gulotta LV. A Comprehensive Enhanced Recovery Pathway for Rotator Cuff Surgery Reduces Pain, Opioid Use, and Side Effects. Clin Orthop Relat Res. 2021 Aug 1;479(8):1740-1751. doi: 10.1097/CORR.0000000000001684. PMID 33720071

RESULTS

PARTICIPANT FLOW:
Groups:
- After Group: We plan to have 70 patients studied after initiation of a pathway.
  Pathway: The study team emphasizes that all components of the pathway are considered standard of care at this institution. The objective of this study is to ensure that the study patients assigned to the pathway will receive these standard of care components.
Period: Overall Study
Arm/Group | Before Group | After Group
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Before Group | After Group | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12) | 59 (10) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 42 | 38 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 66 | 69 | 135
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 62 | 59 | 121
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140
ASA Level [Count of Participants; unit: Participants] — The ASA Physical Status Classification System has been in use for over 60 years. The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. The classification system alone does not predict the perioperative risks, but used with other factors (eg, type of surgery, frailty, level of deconditioning), it can be helpful in predicting perioperative risks. A lower classification is a better "healthier" individual.
  ref: https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system
  Participants
    ASA I | 17 | 12 | 29
    ASA II | 51 | 53 | 104
    ASA III | 2 | 5 | 7
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (5.1) | 28.2 (4.2) | 28.0 (4.7)
Procedure Time [Mean (Standard Deviation); unit: minutes] | 47 (16) | 57 (18) | 52 (18)
Rotator Cuff Repair Performed [Count of Participants; unit: Participants] | 59 | 64 | 123

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome - Worst NRS With Movement
Description: worst NRS with movement. A lower score is a better outcome. The score range is between 0 and 10.
Time Frame: 0-48 hours after block placement
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 70 | 70
score on a scale
  Post-Op Day 1 | 5.6 (3) | 3.3 (3.1)
  Post-Op Day 2 | 6.1 (2.7) | 6.4 (2.5)

2. Secondary Outcome: Total Opioid Use
Description: The total opioid consumption measured in morphine milligram equivalents (MME).
  Although recorded at different time points, the total MME per patient was calculated.
Time Frame: Post Op Days 1,2,7,14
Population: some patients were lost to follow up.
Measure: Median (Inter-Quartile Range); unit: morphine equivalent units (mg)
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 70 | 70
morphine equivalent units (mg)
  0-24 hours | 15 [7.5 to 30] | 0 [0 to 7.5]
  24-48 hours: number analyzed (Participants) | 55 | 50
  24-48 hours | 22.5 [15 to 45] | 15 [7.5 to 30]
  POD7: number analyzed (Participants) | 55 | 64
  POD7 | 0 [0 to 7.5] | 0 [0 to 0]
  POD14: number analyzed (Participants) | 49 | 56
  POD14 | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Patient Satisfaction With Pain Management
Description: Measures the patient's satisfaction with their pain management on a scale of 0-10. A higher score is a better outcome.
Time Frame: Post Op Days 1,2,7,14
Population: Some patients were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 70 | 70
score on a scale
  POD0: number analyzed (Participants) | 69 | 70
  POD0 | 9.6 (1.4) | 9.5 (1.6)
  POD1: number analyzed (Participants) | 62 | 63
  POD1 | 8.2 (2.5) | 9.2 (1.7)
  POD2: number analyzed (Participants) | 60 | 63
  POD2 | 8.6 (1.6) | 8.8 (1.8)
  POD7: number analyzed (Participants) | 56 | 64
  POD7 | 8.7 (1.5) | 9.1 (1.7)
  POD14: number analyzed (Participants) | 51 | 58
  POD14 | 9 (1.3) | 9.1 (1.7)

4. Secondary Outcome: Pain Score at Rest
Description: a NRS score on a scale from 0 to 10. 0 means no pain and 10 is the worst pain imaginable. A lower score is a better outcome.
Time Frame: Post Op Days 1,2,7,14
Measure: Mean (Standard Deviation); unit: score on a scale of
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 70 | 70
score on a scale of
  Post-Op Day 1 | 4.0 (2.9) | 1.9 (2.3)
  Post-Op Day 2 | 4.2 (2.1) | 4.7 (2.8)
  Post-Op Day 7 | 2.3 (2.1) | 3 (2.4)
  Post-Op Day 14 | 2.2 (1.9) | 1.7 (1.4)

5. Secondary Outcome: Block Duration
Description: Measures the duration of the block from:
  the time the block started to the time the block completely wore off the time the block started to the time the patient first noticed pain the time the block started to the time the patient felt normal sensation
Time Frame: Through Post Op Day 2
Population: Some patients were lost to follow up
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Before Group | After Group
Number analyzed (Participants) | 70 | 70
hours
  Time to first notice pain: number analyzed (Participants) | 65 | 50
  Time to first notice pain | 21.1 [13.9 to 23.6] | 25.4 [22.8 to 27.8]
  Time to block start to wear off: number analyzed (Participants) | 67 | 50
  Time to block start to wear off | 20.1 [13.9 to 23.4] | 23.2 [18.3 to 26.9]
  Time to block to completely wear off: number analyzed (Participants) | 65 | 65
  Time to block to completely wear off | 22.7 [17.3 to 24.6] | 28.4 [24.9 to 33.1]
  Time to normal sensation: number analyzed (Participants) | 62 | 61
  Time to normal sensation | 22.8 [17.7 to 26] | 28.6 [25.1 to 36.7]

ADVERSE EVENTS:
Time Frame: Up to postoperative day 14.
Description: This was an observational study so no adverse events were reported. Only post-operative complications were collected.
Arm/Group | Before Group | After Group
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT03717753/Prot_SAP_000.pdf